CLINICAL TRIAL: NCT04380129
Title: A Randomized Clinical Trial Investigating the Effect of the Music Therapy Model "The Bonny Method of Guided Imagery and Music (GIM)" on Patients Suffering From Rheumatoid Arthritis With Chronic Pain
Brief Title: Music Therapy Model "The Bonny Method of Guided Imagery and Music" on Patients With Rheumatoid Arthritis
Acronym: GIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/4ης/11-3-2020
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis; Quality of Life; Chronic Pain
Keywords: Rheumatoid Arthritis; GIM Bonny Method model
MeSH Terms: conditions — Arthritis, Rheumatoid; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Μusic therapy-conversation sessions (Experimental)
  Interventions: Other: Music therapy-conversation sessions
- Music listening (Active Comparator)
  Interventions: Other: Music Listening

INTERVENTIONS:
Other: Music therapy-conversation sessions — The intervention will be performed four times per patient at a frequency once weekly. An effort shall be made to ensure that each treatment is exactly seven days from the previous one within ± one day. The musical hearing will include Helen Bonny's program "Caring", which is proposed by the author of this Music therapy model as the most suitable for patients with chronic and severe pain. The program is as follows:
  * Haydn - Cello Konzert in C, Adagio
  * Dvorak - Serenade in E-Dur, Larghetto
  * Warlock - Capriol Suite, Pieds en I'air
  Other Names: GIM Bonny Method
  Arms: Μusic therapy-conversation sessions
Other: Music Listening — Music Listening to Helen Bonny's programme.
  Arms: Music listening

SUMMARY:
The aim of this study is to investigate the effect of music therapy and in particular of the model "The Bonny Method of Guided Imagery and Music (GIM)" in patients with rheumatoid arthritis (RA) in relation to both chronic pain relief and other psychosocial parameters, as well as the effect of the method on caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis (RA)
* Over 18 years of age

Exclusion Criteria:

•None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Impact of the Bonny Method of Guided Imagery and Music (GIM) on relief of chronic pain from rheumatoid arthritis | 3 years
  The Wong-Baker Face Scale will be used to assess the pain with a simultaneous visual, numeric and functional analog display of the pain the patient is experiencing at the time of the interview. The scale depicts a series of six (6) face faces. The 6 faces are given the following marks:
  * 0 no pain
  * 2 slight pain not affecting certain activities
  * 4 slight pain affecting certain activities
  * 6 moderate pain that does not affect certain activities (such as telephone, TV, reading etc)
  * 8 severe pain affecting certain activities (such as telephone, TV, reading etc)
  * 10 intolerable pain that does not even allow for simple voice communication
The SF-36 questionnaire | 3 years
  The SF-36 questionnaire, simultaneous recording of physical and mental health status of patients will be performed.
The effect of GIM Bonny Method model on the emotional status of careers | 3 years
  The Barthel scale has been used worldwide since it was created in 1965. It is a balanced instrument for scoring basic mobility, self-care and restraint activities, and has 10 thematic areas. The overall score varies from 0 to 100, indicating full dependency and full autonomy, respectively. To be considered autonomous, the patient should not seek human assistance in any of the activities rated. Scale of self-service assessment - Barthel scale
The effect of GIM Bonny Method model on the careers and their relationship with patients both during the intervention period and three months after the first interview | 3 years
  The Zarit Burden Interview (ZBI) questionnaire was created to measure the burden on careers. It consists of 22 questions. The scale score varies from 0-88 and the smaller the score, the smaller the charge.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Larissa, Department of Anesthesiology, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alamanos Y, Drosos AA. Epidemiology of adult rheumatoid arthritis. Autoimmun Rev. 2005 Mar;4(3):130-6. doi: 10.1016/j.autrev.2004.09.002. PMID 15823498
- [Background] Anagnostopoulos F, Niakas D, Pappa E. Construct validation of the Greek SF-36 Health Survey. Qual Life Res. 2005 Oct;14(8):1959-65. doi: 10.1007/s11136-005-3866-8. PMID 16155784
- [Background] Andrianakos A, Trontzas P, Christoyannis F, Kaskani E, Nikolia Z, Tavaniotou E, Georgountzos A, Krachtis P; ESORDIG Study Group. Prevalence and management of rheumatoid arthritis in the general population of Greece--the ESORDIG study. Rheumatology (Oxford). 2006 Dec;45(12):1549-54. doi: 10.1093/rheumatology/kel140. Epub 2006 May 11. PMID 16690763
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] Coons SJ, Rao S, Keininger DL, Hays RD. A comparative review of generic quality-of-life instruments. Pharmacoeconomics. 2000 Jan;17(1):13-35. doi: 10.2165/00019053-200017010-00002. PMID 10747763
- [Background] Cross M, Smith E, Hoy D, Carmona L, Wolfe F, Vos T, Williams B, Gabriel S, Lassere M, Johns N, Buchbinder R, Woolf A, March L. The global burden of rheumatoid arthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1316-22. doi: 10.1136/annrheumdis-2013-204627. Epub 2014 Feb 18. PMID 24550173
- [Background] Dorman PJ, Dennis M, Sandercock P. How do scores on the EuroQol relate to scores on the SF-36 after stroke? Stroke. 1999 Oct;30(10):2146-51. doi: 10.1161/01.str.30.10.2146. PMID 10512920
- [Background] Elliott AM, Smith BH, Hannaford PC, Smith WC, Chambers WA. The course of chronic pain in the community: results of a 4-year follow-up study. Pain. 2002 Sep;99(1-2):299-307. doi: 10.1016/s0304-3959(02)00138-0. PMID 12237208
- [Background] Fishman B, Pasternak S, Wallenstein SL, Houde RW, Holland JC, Foley KM. The Memorial Pain Assessment Card. A valid instrument for the evaluation of cancer pain. Cancer. 1987 Sep 1;60(5):1151-8. doi: 10.1002/1097-0142(19870901)60:53.0.co;2-g. PMID 3300951
- [Background] Gallagher RM. Primary care and pain medicine. A community solution to the public health problem of chronic pain. Med Clin North Am. 1999 May;83(3):555-83, v. doi: 10.1016/s0025-7125(05)70124-3. PMID 10386115
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Jenkinson C, Wright L, Coulter A. Criterion validity and reliability of the SF-36 in a population sample. Qual Life Res. 1994 Feb;3(1):7-12. doi: 10.1007/BF00647843. PMID 8142947
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Mathias SD, Colwell HH, Miller DP, Moreland LW, Buatti M, Wanke L. Health-related quality of life and functional status of patients with rheumatoid arthritis randomly assigned to receive etanercept or placebo. Clin Ther. 2000 Jan;22(1):128-39. doi: 10.1016/s0149-2918(00)87984-9. PMID 10688396
- [Background] das Chagas Medeiros MM, Ferraz MB, Quaresma MR. The effect of rheumatoid arthritis on the quality of life of primary caregivers. J Rheumatol. 2000 Jan;27(1):76-83. PMID 10648021
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Background] Minnock P, Fitzgerald O, Bresnihan B. Quality of life, social support, and knowledge of disease in women with rheumatoid arthritis. Arthritis Rheum. 2003 Apr 15;49(2):221-7. doi: 10.1002/art.11001. PMID 12687514
- [Background] Pappa E, Kontodimopoulos N, Niakas D. Validating and norming of the Greek SF-36 Health Survey. Qual Life Res. 2005 Jun;14(5):1433-8. doi: 10.1007/s11136-004-6014-y. PMID 16047519
- [Background] Sokoll KB, Helliwell PS. Comparison of disability and quality of life in rheumatoid and psoriatic arthritis. J Rheumatol. 2001 Aug;28(8):1842-6. PMID 11508587
- [Background] Stavem K, Lossius MI, Kvien TK, Guldvog B. The health-related quality of life of patients with epilepsy compared with angina pectoris, rheumatoid arthritis, asthma and chronic obstructive pulmonary disease. Qual Life Res. 2000;9(7):865-71. doi: 10.1023/a:1008993821253. PMID 11297029
- [Background] Symmons DP, Barrett EM, Bankhead CR, Scott DG, Silman AJ. The incidence of rheumatoid arthritis in the United Kingdom: results from the Norfolk Arthritis Register. Br J Rheumatol. 1994 Aug;33(8):735-9. doi: 10.1093/rheumatology/33.8.735. PMID 8055200
- [Background] van der Woude D, Houwing-Duistermaat JJ, Toes RE, Huizinga TW, Thomson W, Worthington J, van der Helm-van Mil AH, de Vries RR. Quantitative heritability of anti-citrullinated protein antibody-positive and anti-citrullinated protein antibody-negative rheumatoid arthritis. Arthritis Rheum. 2009 Apr;60(4):916-23. doi: 10.1002/art.24385. PMID 19333951
- [Background] Wild CP. Complementing the genome with an "exposome": the outstanding challenge of environmental exposure measurement in molecular epidemiology. Cancer Epidemiol Biomarkers Prev. 2005 Aug;14(8):1847-50. doi: 10.1158/1055-9965.EPI-05-0456. No abstract available. PMID 16103423
- [Background] Thompson C. The nursing assessment of the patient with cardiac pain on the coronary care unit. Intensive Care Nurs. 1989 Dec;5(4):147-54. doi: 10.1016/0266-612x(89)90002-3. PMID 2621341
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Melzack R, Torgerson WS. On the language of pain. Anesthesiology. 1971 Jan;34(1):50-9. doi: 10.1097/00000542-197101000-00017. No abstract available. PMID 4924784
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Background] Doran MF, Pond GR, Crowson CS, O'Fallon WM, Gabriel SE. Trends in incidence and mortality in rheumatoid arthritis in Rochester, Minnesota, over a forty-year period. Arthritis Rheum. 2002 Mar;46(3):625-31. doi: 10.1002/art.509. PMID 11920397
- [Background] Deschamps M, Band PR, Coldman AJ. Assessment of adult cancer pain: shortcomings of current methods. Pain. 1988 Feb;32(2):133-139. doi: 10.1016/0304-3959(88)90061-9. PMID 3283659